CLINICAL TRIAL: NCT07095543
Title: Feasibility, Implementation, and Efficacy of a Plant-based Online Weight Loss Through Education and Resources Program and Study (POWER Study)
Brief Title: Plant-Based Online Weight Loss Through Education and Resources Program and Study
Acronym: POWER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00087270
Record Dates: First submitted 2025-07-15; First posted 2025-07-31 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes; Overweight and Obese Adults
Keywords: Plant-based diet; Vegan diet; type 2 diabetes; Weight loss; Overweight; Obesity; Cholesterol
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Weight Loss; Obesity | interventions — Diet, Fat-Restricted; Diet, Vegan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-fat, vegan diet (Experimental): All participants will be asked to follow a low-fat vegan diet. There are no other study arms or control group.
  Interventions: Behavioral: Low-fat, vegan diet

INTERVENTIONS:
Behavioral: Low-fat, vegan diet — All participants will be asked to follow a low-fat vegan diet for the duration of the study. Participants will attend weekly classes where they we receive education and support.

SUMMARY:
This is an interventional study that will evaluate the feasibility, implementation, and efficacy of an online, 12-week, plant-based, nutrition education program in a community setting. Participants will meet with a physician and a registered dietitian once a week to learn about a plant-based diet and receive support and practical help in making the dietary changes. Body composition, blood sugar control, cholesterol levels, and food costs will be measured at the start and end of the study.

DETAILED DESCRIPTION:
This is an interventional study that will evaluate the feasibility, implementation, and efficacy of an online, 12-week, plant-based, nutrition education program in a community setting. Participants will participate in weekly physician- and dietitian-lead group classes and will receive education about a plant-based diet as well as support and practical tips for implementing the dietary changes. Participants will receive baseline and 12 week assessments including a DXA scan to assess body composition, HbA1c, lipid panel, and a food cost analysis.

ELIGIBILITY:
Inclusion Criteria:

* U.S. men and women meeting the age of majority, defined as follows:

Age 19 or older in Nebraska and Alabama. Age 21 or older in Puerto Rico. Age 18 or older in all other states.

* Able and willing to travel to Washington DC for a dual-energy х-rау absorptiometry (DXA) scans before and after the program.
* Able and willing to complete laboratory assessments at a local LabCorp facility before and after the program.
* Able and willing to participate in all components of the study.
* BMI of 25 or more (23 or more in persons of Asian origin).
* Access to the internet.
* English fluency.

Exclusion Criteria:

* Use of recreational drugs in the past 6 months.
* Pregnancy or intention to become pregnant during the study period, as verified by self-report.
* Unstable medical or psychiatric illness.
* Inability to maintain medication regimen as prescribed by personal healthcare provider.
* Current or expected use of any weight loss medication during the study period, including but not limited to, glucagon-like peptide-1 (GLP-1) receptor agonists and combination GLP-1 receptor/glucose-dependent insulinotropic polypeptide (GIP) agonists.
* Use of any weight loss medication within the 12 months preceding the study period, including but not limited to, glucagon-like peptide-1 (GLP-1) receptor agonists and combination GLP-1 receptor/glucose-dependent insulinotropic polypeptide (GIP) agonists.
* Body weight greater than 182 kg.
* Current diagnosis of eating disorder.
* Intention to follow another weight loss method during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
The feasibility of an online plant-based weight loss program in the community setting. | From baseline to the end of the intervention at 12 weeks.
  Feasibility will be assessed by the number of total participants that enroll in the program and complete both baseline and final assessments.

SECONDARY OUTCOMES:
Changes in glycated hemoglobin. | From baseline to the end of the intervention at 12 weeks.
  A1c will be measured using standard methods.
Changes in total and LDL cholesterol levels. | From baseline to the end of the intervention at 12 weeks.
  Total and LDL cholesterol levels will be measured using standard methods.
Changes in body composition. | From baseline to the end of the intervention at 12 weeks.
  Body composition will be measured by dual energy x-ray absorptometry (Lunar iDXA, GE Healthcare; Madison, WI) with Encore® 2005 v.9.15.010 software. The iDXA can measure body composition with low x-ray exposure and short scanning time. The iDXA unit will be calibrated daily using the GE Lunar calibration phantom, and a trained operator will perform all scans following standard protocol for participant positioning. The iDXA is equipped with the CoreScan module (GE Healthcare, Madison, WI), which can also provide an estimate of visceral adipose tissue volume and mass.
Food costs of a baseline diet and a low-fat plant-based diet. | From baseline to the end of the intervention at 12 weeks.
  Study participants will be asked to provide a food consumption record of three consecutive days (including two weekdays and one weekend day). Participants will be asked to include the specific brands, portions, names of retailers and restaurants where the food was purchased. A study team member will review the food record with the participants. We will then calculate the total cost of the food consumed during the 3-day period using cost data from the retailers' and restaurants' websites or by calling the specific restaurants and retailers.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kahleova H, Sutton M, Maracine C, Nichols D, Monsivais P, Holubkov R, Barnard ND. Food Costs of a Low-Fat Vegan Diet vs a Mediterranean Diet: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2445784. doi: 10.1001/jamanetworkopen.2024.45784. PMID 39556398
- [Background] Kahleova H, Sutton M, Maracine C, Nichols D, Monsivais P, Holubkov R, Barnard ND. Vegan Diet and Food Costs Among Adults With Overweight: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Sep 5;6(9):e2332106. doi: 10.1001/jamanetworkopen.2023.32106. PMID 37669055
- [Background] Stanford J, Zuck M, Stefoska-Needham A, Charlton K, Lambert K. Acceptability of Plant-Based Diets for People with Chronic Kidney Disease: Perspectives of Renal Dietitians. Nutrients. 2022 Jan 4;14(1):216. doi: 10.3390/nu14010216. PMID 35011091
- [Background] Barnard ND, Gloede L, Cohen J, Jenkins DJ, Turner-McGrievy G, Green AA, Ferdowsian H. A low-fat vegan diet elicits greater macronutrient changes, but is comparable in adherence and acceptability, compared with a more conventional diabetes diet among individuals with type 2 diabetes. J Am Diet Assoc. 2009 Feb;109(2):263-72. doi: 10.1016/j.jada.2008.10.049. PMID 19167953
- [Background] Emamat H, Jamshidi A, Farhadi A, Ghalandari H, Ghasemi M, Tangestani H. The association between the visceral to subcutaneous abdominal fat ratio and the risk of cardiovascular diseases: a systematic review. BMC Public Health. 2024 Jul 9;24(1):1827. doi: 10.1186/s12889-024-19358-0. PMID 38982435
- [Background] Yokoyama Y, Levin SM, Barnard ND. Association between plant-based diets and plasma lipids: a systematic review and meta-analysis. Nutr Rev. 2017 Sep 1;75(9):683-698. doi: 10.1093/nutrit/nux030. PMID 28938794
- [Background] Kahleova H, Petersen KF, Shulman GI, Alwarith J, Rembert E, Tura A, Hill M, Holubkov R, Barnard ND. Effect of a Low-Fat Vegan Diet on Body Weight, Insulin Sensitivity, Postprandial Metabolism, and Intramyocellular and Hepatocellular Lipid Levels in Overweight Adults: A Randomized Clinical Trial. JAMA Netw Open. 2020 Nov 2;3(11):e2025454. doi: 10.1001/jamanetworkopen.2020.25454. PMID 33252690
- [Background] Kahleova H, Tura A, Hill M, Holubkov R, Barnard ND. A Plant-Based Dietary Intervention Improves Beta-Cell Function and Insulin Resistance in Overweight Adults: A 16-Week Randomized Clinical Trial. Nutrients. 2018 Feb 9;10(2):189. doi: 10.3390/nu10020189. PMID 29425120
- [Background] Campbell TM, Campbell EK, Attia J, Ventura K, Mathews T, Chhabra KH, Blanchard LM, Wixom N, Faniyan TS, Peterson DR, Harrington DK, Wittlin SD. The acute effects of a DASH diet and whole food, plant-based diet on insulin requirements and related cardiometabolic markers in individuals with insulin-treated type 2 diabetes. Diabetes Res Clin Pract. 2023 Aug;202:110814. doi: 10.1016/j.diabres.2023.110814. Epub 2023 Jul 5. PMID 37419391
- [Background] Barnard ND, Cohen J, Jenkins DJ, Turner-McGrievy G, Gloede L, Jaster B, Seidl K, Green AA, Talpers S. A low-fat vegan diet improves glycemic control and cardiovascular risk factors in a randomized clinical trial in individuals with type 2 diabetes. Diabetes Care. 2006 Aug;29(8):1777-83. doi: 10.2337/dc06-0606. PMID 16873779
- [Background] Gwira JA, Fryar CD, Gu Q. Prevalence of Total, Diagnosed, and Undiagnosed Diabetes in Adults: United States, August 2021-August 2023. NCHS Data Brief. 2024 Nov;(516):CS354814. doi: 10.15620/cdc/165794. PMID 40085919
- [Background] Barnard ND, Alwarith J, Rembert E, Brandon L, Nguyen M, Goergen A, Horne T, do Nascimento GF, Lakkadi K, Tura A, Holubkov R, Kahleova H. A Mediterranean Diet and Low-Fat Vegan Diet to Improve Body Weight and Cardiometabolic Risk Factors: A Randomized, Cross-over Trial. J Am Nutr Assoc. 2022 Feb;41(2):127-139. doi: 10.1080/07315724.2020.1869625. Epub 2021 Feb 5. PMID 33544066
- [Background] Global BMI Mortality Collaboration, Di Angelantonio E, Bhupathiraju ShN, Wormser D, Gao P, Kaptoge S, Berrington de Gonzalez A, Cairns BJ, Huxley R, Jackson ChL, Joshy G, Lewington S, Manson JE, Murphy N, Patel AV, Samet JM, Woodward M, Zheng W, Zhou M, Bansal N, Barricarte A, Carter B, Cerhan JR, Smith GD, Fang X, Franco OH, Green J, Halsey J, Hildebrand JS, Jung KJ, Korda RJ, McLerran DF, Moore SC, O'Keeffe LM, Paige E, Ramond A, Reeves GK, Rolland B, Sacerdote C, Sattar N, Sofianopoulou E, Stevens J, Thun M, Ueshima H, Yang L, Yun YD, Willeit P, Banks E, Beral V, Chen Zh, Gapstur SM, Gunter MJ, Hartge P, Jee SH, Lam TH, Peto R, Potter JD, Willett WC, Thompson SG, Danesh J, Hu FB. Body-mass index and all-cause mortality: individual-participant-data meta-analysis of 239 prospective studies in four continents. Lancet. 2016 Aug 20;388(10046):776-86. doi: 10.1016/S0140-6736(16)30175-1. Epub 2016 Jul 13. PMID 27423262
- [Background] Kivimaki M, Kuosma E, Ferrie JE, Luukkonen R, Nyberg ST, Alfredsson L, Batty GD, Brunner EJ, Fransson E, Goldberg M, Knutsson A, Koskenvuo M, Nordin M, Oksanen T, Pentti J, Rugulies R, Shipley MJ, Singh-Manoux A, Steptoe A, Suominen SB, Theorell T, Vahtera J, Virtanen M, Westerholm P, Westerlund H, Zins M, Hamer M, Bell JA, Tabak AG, Jokela M. Overweight, obesity, and risk of cardiometabolic multimorbidity: pooled analysis of individual-level data for 120 813 adults from 16 cohort studies from the USA and Europe. Lancet Public Health. 2017 May 19;2(6):e277-e285. doi: 10.1016/S2468-2667(17)30074-9. eCollection 2017 Jun. PMID 28626830
- [Background] Emmerich SD, Fryar CD, Stierman B, Ogden CL. Obesity and Severe Obesity Prevalence in Adults: United States, August 2021-August 2023. NCHS Data Brief. 2024 Sep;(508):10.15620/cdc/159281. doi: 10.15620/cdc/159281. PMID 39808758